CLINICAL TRIAL: NCT00006096
Title: A Randomized Study of Adjuvant Radiation Treatment Versus Radiation and Chemotherapy in Patients With Vulvar Cancer and Involved Nodes
Brief Title: Radiation Therapy With or Without Cisplatin in Treating Patients With Stage I, Stage II, or Stage III Cancer of the Vulva
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068103; GOG-0185
Record Dates: First submitted 2000-08-03; First posted 2003-09-03 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2007-06

CONDITIONS: Vulvar Cancer
Keywords: stage I vulvar cancer; stage II vulvar cancer; stage III vulvar cancer; stage IVB vulvar cancer; squamous cell carcinoma of the vulva
MeSH Terms: conditions — Vulvar Neoplasms | interventions — Cisplatin; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if radiation therapy combined with chemotherapy kills more tumor cells than radiation therapy alone in treating cancer of the vulva.

PURPOSE: Randomized phase III trial to determine the effectiveness of radiation therapy with or without cisplatin in treating patients who have stage I, stage II, or stage III cancer of the vulva.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the recurrence-free interval and survival in patients with stage I, II, III, or IVA squamous cell carcinoma of the vulva with involved inguinal lymph nodes treated with adjuvant radiotherapy with or without cisplatin.
* Compare the toxicity of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to primary surgical resection (yes vs no) and node status (N1 vs N2). Patients are randomized to one of two treatment arms.

* Arm I: Patients undergo radiotherapy 5 days a week for 6 weeks.
* Arm II: Patients undergo radiotherapy as in arm I. Patients also receive cisplatin IV over 1 hour on days 1, 8, 15, 22, 29, and 36.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 250 patients will be accrued for this study within 4.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage I, II, III, or IVA squamous cell carcinoma of the vulva amenable to curative treatment with surgery, radiotherapy, or both

  * At least 1 positive inguinal and/or femoral lymph node
  * No inoperable (fixed or ulcerating) groin nodes
  * Must not require resection of urethra or anal sphincter to achieve negative margins
* Must have undergone vulvar biopsy and bilateral inguinal/femoral lymph node dissection within 8 weeks of randomization
* No metastatic disease

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* GOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Granulocyte count at least 1,500/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times normal
* SGOT no greater than 3 times normal
* Alkaline phosphatase no greater than 3 times normal

Renal:

* Creatinine no greater than 2.0 mg/dL

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other prior invasive malignancy within the past 5 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy

Surgery:

* See Disease Characteristics
* No more than 8 weeks since prior surgery

Other:

* No prior therapy for another malignancy that would preclude study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-03; Primary Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gillian M. Thomas, BSc, MD, FRCPC, FRCR (Hon), Study Chair — GlaxoSmithKline
Locations (30):
- United States (28):
  - Community Hospital of Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of Colorado Cancer Center, Denver, Colorado
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Tufts University School of Medicine, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - Cancer Center of Albany Medical Center, Albany, New York
  - Schneider Children's Hospital at North Shore, Manhasset, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Brookview Research, Inc., Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - M.D. Anderson CCOP Research Base, Houston, Texas
  - Fletcher Allen Health Care - Medical Center Campus, Burlington, Vermont
  - Tacoma General Hospital, Tacoma, Washington
- Canada (2):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario